CLINICAL TRIAL: NCT05663775
Title: Prophylactic Oral Mesalamine for the Prevention of Immune-Related Colitis in Patients Treated With Ipilimumab/Nivolumab
Brief Title: Prophylactic Mesalamine to Prevent Colitis Following Treatment With Ipilimumab/Nivolumab (Ipi/Nivo)
Acronym: IMPACT 1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT-0007
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Immune-related Adverse Event; Diarrhea; Advanced Melanoma; Advanced Rectal Carcinoma
MeSH Terms: conditions — Diarrhea | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prophylactic Mesalamine in combination of Immunotherapy (Nivolumab/Ipilimumab) (Experimental): Participants will receive 500mg of Mesalamine QID (four times a day) in combination with standard of care Immunotherapy
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine — Mesalamine, also known as 5-aminosalicylic acid (5-ASA)
  Other Names: Salofalk

SUMMARY:
The study team's principal interest is to address the question, "Will prophylactic treatment with mesalamine reduce the incidence and severity of immune-related diarrhea occurring secondarily to treatment with ipi/nivo?"

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients with histologically confirmed, unresectable stage III or IV malignant melanoma.
3. Patients must be capable of providing consent to enrolment and treatment.
4. Patients with a performance status of ECOG 0-224 will be eligible for enrolment (see appendix16.1).
5. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
6. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 30 days after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   -Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
7. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 30 days after the last dose of study drug.
8. Male patients should agree to not donate sperm during the study and for a period of at least 30 days after last dose of study drug
9. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.

   * The following adequate organ function laboratory values must be met:

Hematological:

* Absolute neutrophil count (ANC) >1.5 x109/L
* Platelet count >100 x109/L
* Hemoglobin >9 g/dL (may have been transfused)

Renal:

o Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)

Hepatic:

* Total serum bilirubin <2x ULN
* AST and ALT <2.5x ULN (or ≤ 5 x ULN for subjects with documented metastatic disease to the liver)

Exclusion Criteria:

1. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
2. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
3. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAE v5 Grade ≥ 3).
4. Other severe acute or chronic medical conditions or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related Diarrhea | Diarrhea (incidence) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Diarrhea will be graded according to parameters described within the CTCAE v5.0.
Severity of Treatment Related Diarrhea | Diarrhea (severity) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Diarrhea will be graded according to parameters described within the CTCAE v5.0.
Causality of Treatment Related Diarrhea | Diarrhea (causality) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Diarrhea will be graded according to parameters described within the CTCAE v5.0. The cause for diarrhea (treatment-related or not) will be assessed by the treating physician/investigator.

SECONDARY OUTCOMES:
Incidence of all IR-AEs (diarrheal and non-diarrheal, all grades) | IR-AEs (incidence and severity, as well as causality) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks)and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Adverse events deemed immune-related will be graded according to parameters described within the CTCAE v5.0. The treating physician/investigator will be responsible for determining whether or not an adverse event is immune-related.
Incidence of IR-AEs ≥ grade 2 | IR-AEs that are greater than grade 2 (incidence and severity, as well as causality) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Adverse events deemed immune-related will be graded according to parameters described within the CTCAE v5.0. The treating physician/investigator will be responsible for determining whether or not an adverse event is immune-related.
Times to onset and resolution of IR-AEs | IR-AEs (incidence and severity, as well as causality) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  Adverse events deemed immune-related will be graded according to parameters described within the CTCAE v5.0. The treating physician/investigator will be responsible for determining whether or not an adverse event is immune-related. The onset of IR-AEs shall be defined as that point in time when a study participant first described signs or symptoms indicative of an IR-AE. Resolution of an IR-AE shall be defined as that point in time when an IR-AE resolves, or in the case where a particular sign/symptom was present prior to study enrolment, the individual participant's baseline.
Requirement for immunosuppressive (steroid and non-steroid) medications to manage IR-AEs | Concomitant Medications will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  The use of steroidal and non-steroidal immunosuppressive therapies will be analyzed during a participant's time on study. The designation of a particular therapy as "immunosuppressive," including whether or not the therapy may be classified as steroidal or non-steroidal will be performed by the treating physician/investigator. Information regarding specific therapy(s) prescribed, as well as duration of said therapy will be collected.
Frequency of IR-AEs leading to treatment discontinuation | IR-AEs (incidence and severity, as well as causality) will be assessed at each Screening, Cycle 1-4 (each cycle is 3 weeks) and throughout the post treatment follow-up (12, 18 and 24 weeks)
  During collection of data regarding incidence/severity of IR-AEs, information regarding whether or not treatment was held (dose-limiting) or permanently discontinued (treatment-limiting) will be collected. As described above, grading of IR-AEs will be in accordance with CTCAE guidance, and assignment of causality will be the responsibility of the treating physician/investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided